CLINICAL TRIAL: NCT06828653
Title: Feasibility RCT Evaluating Digitally and Traditionally Produced Ankle Foot Orthoses for Individuals With Impaired Lower Limb Function
Brief Title: Comparing Digitally and Traditionally Made Ankle Foot Orthoses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 703
Record Dates: First submitted 2025-02-03; First posted 2025-02-14 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Flaccid Paresis; Spastic Paresis; Cerebral Palsy; Stroke; Spinal Cord Injury; Spina Bifida; Traumatic Peripheral Nerve Injury
Keywords: Ankle foot orthosis; ankle foot orthoses; digital ankle foot orthoses; digital technology; 3D scanning; 3D printing; randomized control trial
MeSH Terms: conditions — Cerebral Palsy; Stroke; Spinal Cord Injuries; Spinal Dysraphism

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: Traditional AFO(s) wear first; Part B: Traditional AFO(s) wear (Active Comparator): Participants wear traditionally produced AFO(s) for 3 weeks, and will then crossover to wear digital AFO(s) for another 3 weeks. In Part B of the study, participants will wear traditional AFO(s) for 8 weeks.
  Interventions: Device: Part A First Wear Period: Traditional AFO(s); Device: Part A Second Wear Period: Digital AFO(s); Device: Part B Long-term Evaluation Period: Traditional AFO(s)
- Part A: Digital AFO(s) wear first; Part B: Digital AFO(s) wear (Experimental): Participants wear digitally produced AFO(s) for 3 weeks, and will then crossover to wear traditional AFO(s) for another 3 weeks. In Part B of the study, participants will wear digital AFO(s) for 8 weeks.
  Interventions: Device: Part A First Wear Period: Digital AFO(s); Device: Part A Second Wear Period: Traditional AFO(s); Device: Part B Long-term Evaluation Period: Digital AFO(s)
- Part A: Traditional AFO(s) wear first; Part B: Digital AFO(s) wear (Active Comparator): Participants wear traditionally produced AFO(s) for 3 weeks, and will then crossover to wear digital AFO(s) for another 3 weeks. In Part B of the study, participants will wear digital AFO(s) for 8 weeks.
  Interventions: Device: Part A First Wear Period: Traditional AFO(s); Device: Part A Second Wear Period: Digital AFO(s); Device: Part B Long-term Evaluation Period: Digital AFO(s)
- Part A: Digital AFO(s) wear first; Part B: Traditional AFO(s) wear (Active Comparator): Participants wear digitally produced AFO(s) for 3 weeks, and will then crossover to wear traditional AFO(s) for another 3 weeks. In Part B of the study, participants will wear traditional AFO(s) for 8 weeks.
  Interventions: Device: Part A First Wear Period: Digital AFO(s); Device: Part A Second Wear Period: Traditional AFO(s); Device: Part B Long-term Evaluation Period: Traditional AFO(s)

INTERVENTIONS:
Device: Part A First Wear Period: Traditional AFO(s) — Participants are randomized to wear traditionally produced AFOs during Weeks 1 through 3.
  Arms: Part A: Traditional AFO(s) wear first; Part B: Digital AFO(s) wear; Part A: Traditional AFO(s) wear first; Part B: Traditional AFO(s) wear
Device: Part A First Wear Period: Digital AFO(s) — Participants are randomized to wear digitally produced AFOs during Weeks 1 through 3.
  Arms: Part A: Digital AFO(s) wear first; Part B: Digital AFO(s) wear; Part A: Digital AFO(s) wear first; Part B: Traditional AFO(s) wear
Device: Part A Second Wear Period: Traditional AFO(s) — Participants wear traditionally produced AFOs during Weeks 4 through 6.
  Arms: Part A: Digital AFO(s) wear first; Part B: Digital AFO(s) wear; Part A: Digital AFO(s) wear first; Part B: Traditional AFO(s) wear
Device: Part A Second Wear Period: Digital AFO(s) — Participants wear digitally produced AFOs during Weeks 4 through 6.
  Arms: Part A: Traditional AFO(s) wear first; Part B: Digital AFO(s) wear; Part A: Traditional AFO(s) wear first; Part B: Traditional AFO(s) wear
Device: Part B Long-term Evaluation Period: Traditional AFO(s) — Participants are randomized to wear traditionally produced AFO(s) during Weeks 7 through 14.
  Arms: Part A: Digital AFO(s) wear first; Part B: Traditional AFO(s) wear; Part A: Traditional AFO(s) wear first; Part B: Traditional AFO(s) wear
Device: Part B Long-term Evaluation Period: Digital AFO(s) — Participants are randomized to wear digitally produced AFO(s) during Weeks 7 through 14.
  Arms: Part A: Digital AFO(s) wear first; Part B: Digital AFO(s) wear; Part A: Traditional AFO(s) wear first; Part B: Digital AFO(s) wear

SUMMARY:
The research is being done to compare two methods of creating AFOs: 1. The traditional method, which involves manually creating a mold from a plaster cast of the client's limb. This is time-consuming and labor-intensive; and 2. The newer method uses digital technology, such as 3D scanning and printing, to design and produce the AFOs, potentially making the process faster and less costly. We want to know whether AFOs made using digital technology can provide the same clinical benefits as those made traditionally.

DETAILED DESCRIPTION:
This study is designed to compare two methods of creating ankle-foot orthoses (AFOs), which are devices used to support the lower limbs in people with mobility impairments due to conditions like stroke or cerebral palsy. The traditional method involves manually creating a mold from a plaster cast of the patient's limb, which is time-consuming and labor-intensive. The new method uses digital technology, such as 3D scanning and printing, to design and produce the AFOs, potentially making the process faster and less costly.

The purpose of the study is to test whether AFOs made using digital technology can provide the same clinical benefits as those made traditionally, but with greater efficiency and at a lower cost. The research will gather data on patient satisfaction, the functionality of the AFOs, and the costs associated with each method. This will help determine if the digital method can be a viable alternative to traditional AFO production, potentially leading to better patient care and reduced healthcare costs.

The study poses the overarching research question: Can digitally produced ankle-foot orthoses (AFOs) achieve similar positive clinical outcomes to traditionally fabricated AFOs while being more efficient and cost-effective? The primary objective of this feasibility study is to inform the design of a larger randomized controlled trial (RCT) that will comprehensively address this question.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged 8 years or older.
* Participants should have either flaccid or spastic paresis resulting from conditions such as cerebral palsy, stroke, spinal cord injury, spina bifida, or traumatic peripheral nerve injury, leading to lower limb mobility impairments.
* Participants must require a custom articulating, rigid, or energy storage and return (ESR) AFO to improve physical function for one or both sides (unilateral or bilateral).
* Participants must be able to ambulate independently, though the use of gait aids is permitted.
* Participants must be capable of completing questionnaires with no more than orienting guidance.
* Participants must meet the requirements to have their AFO funded by the Assistive Devices Program (ADP).

Exclusion Criteria:

* Clients for whom the primary goal of the AFO includes wound management.
* Those whose AFO is not worn for ambulation.
* Clients with insensate feet or a history of ulcerations.
* First-time AFO users.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) | From the shape capture visit until the end of the study at week 14
  Evaluates patient satisfaction related to assistive technology and services rendered. This questionnaire is commonly used in assessing performance of AFOs and other orthotic devices.

SECONDARY OUTCOMES:
Orthotic Patient-Reported Outcomes - Mobility (OPRO-M) | From Week 1 until Week 6 of the study
  Designed and validated to assess orthotic users' ability to perform activities related to movement, locomotion, and/or postural transitions.
Orthotics Prosthetics User's Survey (OPUS) | From Week 1 until Week 6 of the study
  Assesses function, satisfaction, and quality of life of individuals using orthotic or prosthetic devices. Its Lower Extremity Functional Status component will be used since it pertains specifically to the individual's functional abilities and limitations.
10-metre Walk Test | From the shape capture visit until the end of the study at Week 14
  Timed walk test
Timed Up and Go (TUG) | From the shape capture visit until the end of the study at Week 14
Goal Attainment Scale (GAS) | From the shape capture appointment until the participant receives their devices at Week 1
  Creating biomechanical (alignment/dynamic) goals that AFOs are designed to treat. Will be applied to both types of AFOs. Goal achievement rating will be based on a modification of the GAS 5-level rating system (levels -2 to 0 only) after AFO fitting is complete
AFO Challenge | From the shape capture visit until the end of the study at Week 14
  A new six-item measure that was created by the Holland Bloorview team for this study to capture any functionally important differences in balance linked with AFO type across a spectrum of client abilities.
Orthotist Satisfaction Questionnaire | From the shape capture visit until the end of the crossover period at Week 6
  Evaluate orthotists' satisfaction with the AFO fabrication and fitting process.
Orthotic Patient-Reported Outcomes - Mobility (OPRO-M) | From the shape capture visit until the end of the crossover period at Week 6
  Designed and validated to assess orthotic users' ability to perform activities related to movement, locomotion, and/or postural transitions.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Andrysek, P.Eng, PhD, Principal Investigator — Bloorview Research Institute; Virginia Wright, PT, PhD, Principal Investigator — Bloorview Research Institute
Locations (2):
- Canada (2):
  - Boundless Biomechanical Bracing, Mississauga, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No